CLINICAL TRIAL: NCT03067584
Title: Genetic Study of Familial Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FAMALL2
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: Familial cancer; Genetic predisposition; Heritable disease; Cancer risk; Genome analysis; Genetic modifiers; Next generation sequencing (NGS); Genetic counseling; DNA
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and tumor/tissue for DNA testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Familial aggregation is well recognized in some cancers. Though a number of familial cancer predisposition syndromes have been described, the nature of inherited genetic alterations in patients with a strong history of familial cancer is currently unknown, as is the case with childhood acute lymphoblastic leukemia (ALL).

The investigators are seeking to learn more about what causes leukemia and why some people and families may be at a higher risk of developing this disease. By understanding the origin of the disease, better treatments may be identified for patients with leukemia.

PRIMARY OBJECTIVE: To identify variants in genes that are inherited, have altered gene structure and/or function, and influence the risk of developing acute lymphoblastic leukemia (ALL) and other cancers.

SECONDARY OBJECTIVE: To collect demographic, clinical and laboratory information including detailed family cancer history and response of cancers to therapy for correlation with the primary objective.

DETAILED DESCRIPTION:
This study entails clinical interviews, submission of a peripheral germline blood sample for non-tumor DNA and permission to perform biologic studies on previously stored tumor tissue if applicable and available. Participants diagnosed with cancer at outside institutions will be requested to sign a release form to allow the outside institution to send germline and/or tumor tissue to St Jude if available. For patients who have undergone a stem cell transplant, a buccal swab or saliva sample will be requested (for germline DNA). For patients with active leukemia, non-tumor cells (for germline DNA) may be obtained using a remission blood sample, a skin biopsy (to obtain fibroblasts) or may be purified by fluorescence activated cell sorting of leukemia samples. The skin biopsy will be obtained in participants 18 years of age and older. In participants less than 18 years, the skin biopsy will be accessed only if it was already collected as part of another research protocol or for clinical care.

All patients being considered for enrollment will have a clinical genetics consult by one of the study team members at which time a family history will be taken and information about genomic testing will be introduced. Detailed medical history will be obtained which includes but is not limited to demographics, clinical data including laboratory results, cancer history/diagnosis, treatment outcomes, environmental exposures and cancer risk factors to enable phenotype/genotype correlations.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute lymphoblastic leukemia (ALL) and has a relative also diagnosed with ALL. Note: There is no upper age limit, and the index ALL case does not have to be a patient diagnosed and/or treated at St. Jude.
* Family members of the patient, either affected or unaffected by a malignancy, who are contacted by the patient (or guardian) and agree to participate in the study. Relatives may have been diagnosed with other malignant, genetic or developmental disorders.
* Research participant or legal guardian, as appropriate, must provide informed consent for this protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (proband) with ALL and their relatives with and without ALL.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Identification of novel cancer predisposing genes | Up to 10 years following study activation
  Probands and cancer affected and unaffected relatives from selected families will be sequenced using Whole Genome Sequencing (WGS) or possibly Whole Exome Sequencing (WES) and analyzed to identify new predisposing genetic variants that co-segregate with the tumor phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: John T. Sandlund, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols